CLINICAL TRIAL: NCT00137553
Title: The Efficacy of Re-treatment With Sulfadoxine-pyrimethamine in Children With Recrudescent Malaria in Guinea-Bissau
Brief Title: The Efficacy of Re-treatment With Sulfadoxine-pyrimethamine in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bandim Health Project (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSB-2001-Fansidar
Record Dates: First submitted 2005-08-28; First posted 2005-08-30 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2010-03

CONDITIONS: Malaria, Falciparum
Keywords: Children; malaria; sulfadoxine-pyrimethamine; Guinea-Bissau; treatment
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — fanasil, pyrimethamine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sulfadoxine-pyrimethamine (Fansidar)

SUMMARY:
Children participating in a study evaluating the efficacy of chloroquine and amodiaquine for the treatment of malaria will, if getting malaria during follow-up, be re-treated with sulfadoxine-pyrimethamine (SP) in accordance with the recommendations of the National Malaria Programme.

To compare the actual efficacy of SP with that in 1995 - 1996 we, the investigators of the Bandim Health Project, will visit these children once a week for 5 weeks. A finger prick blood sample will be collected for a malaria test.

Children with malaria during follow-up will be treated according to the guidelines of the Bandim Health Centre.

DETAILED DESCRIPTION:
The Bandim Health Project studies the efficacy of different treatment regimens for malaria in children. If the included children during follow-up get malaria again they are, according to the recommendations of the National Malaria Programme, treated with sulfadoxine-pyrimethamine (SP).

In 1995 - 1996 the efficacy of this re-treatment regimen was evaluated in the same area.

To evaluate if treatment with SP is still efficient we want to follow children included in a study comparing treatment with chloroquine and amodiaquine having recrudescent malaria for 35 days following the re-treatment with SP.

Children with reappearing parasitaemia will be treated with SP. If accepting to participate in this study the children will be visited once a week and a capillary blood sample will be drawn. The blood sample taken on the day of reappearing parasitaemia in the chloroquine/amodiaquine study will be used as the day 0 blood sample in the SP-study.

If the child gets malaria during the follow-up he will be treated according to the guidelines of the Bandim Health Centre. All treatment during follow-up will be free.

ELIGIBILITY:
Inclusion Criteria:

* Malaria symptoms plus positive malaria film
* > 20 parasites per 200 leukocytes
* Treatment failure in a study comparing chloroquine and amodiaquine
* Informed consent

Exclusion Criteria:

* Stated allergy to sulfadoxine and/or pyrimethamine

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60
Dates: Start 2001-05; Study Completion 2004-03

PRIMARY OUTCOMES:
Re-appearing parasitaemia

CONTACTS AND LOCATIONS:
Overall Officials: Peter Aaby, Professor, Study Director — Bandim Health Project
Locations (1):
- Bandim Health Project, Apartado 861, Bissau Region, Guinea-Bissau